CLINICAL TRIAL: NCT06326424
Title: Delirium Identification in Older Patients With Alzheimer's and Other Related Dementias In the Emergency Department Using Wrist Accelerometer Biosensors and Machine Learning
Brief Title: Delirium Identification in Older Patients With Alzheimer's and Other Related Dementias In the Emergency Department
Acronym: DELIRIUM
Status: Recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Lauren Southerland, Associate Professor, Ohio State University
Other Study IDs: 2023H0085
Record Dates: First submitted 2024-03-05; First posted 2024-03-22 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Delirium; Dementia; Hospital Acquired Condition
Keywords: emergency department; delirium; older adults; dementia
MeSH Terms: conditions — Delirium; Dementia; Iatrogenic Disease; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational DELIRIUM cohort: We will follow up to 60 adults 65+ years old with dementia or suspected dementia who are likely to be in the emergency department, observation unit, or hospital for 48 hours. We will follow them for up to 48 hours while they wear an FDA approved biosensor watch and perform delirium checks.
  Interventions: Device: Empatica EmbracePlus

INTERVENTIONS:
Device: Empatica EmbracePlus — wear a biosensor watch to passively collect biosensor data over 48 hours. The EmbracePlus will collect heart rate variability, accelerometry, and electrodermal activity.

SUMMARY:
Delirium is highly prevalent and very bad for patients with dementia. Delirium is a dangerous medical condition that occurs in 6-38% of older Emergency Department patients and 70% of ICU patients. A person who develops delirium in the ED or hospital has a 12 times higher odds of being newly diagnosed with dementia in the next year compared to a similar patient who does not become delirious. Delirium is especially dangerous for persons living with Alzheimer Disease and Related Dementias (AD/ADRD). Persons living with ADRD have an almost 50% chance of developing delirium in the hospital.

Clinicians are bad at recognizing delirium. A recent systematic review led by the Geriatric Emergency Care Applied Research network (NIH funded) found that current delirium screening tools are at most 64% sensitive, meaning that physicians can identify some phenotypes of delirium well, but cannot easily rule out delirium in acutely ill older patients.

The investigators propose integrating wrist biosensors into the emergency management of older adults with dementia. The investigators will monitor heart rate variability, movement, and electrodermal activity (electrical activity of at the level of the skin) to determine if an array of biosensors more sensitive to delirium than current verbal screening tools.

DETAILED DESCRIPTION:
Aim 1: (Patient and Caregiver Acceptability) Collect biosensor data on 60 older adults with dementia in the ED. The study population is any older adult with dementia in the ED who is anticipated to be in the ED or hospital for >4 hours. The investigators will place a wrist biosensor on the dominant hand (unless prohibited by IV placement, in which case the nondominant hand will be used). The investigators will ask questions about acceptability to caregiver (if available) and patient within 4-24 hour mark after biosensor placement. The acceptability questions are derived from the Theoretical Framework of Acceptability Questionnaire.

Study end data will be collected in person prior to discharge, but if unable to be completed before discharge from the hospital, the investigators will call them back at home to complete the final survey about acceptability.

Aim 2: Correlation of biosensor data with delirium phenotype. RA will perform a CAM ICU 7 upon enrollment, and at 24 and 48 hours (or upon discharge, whichever comes first). The investigators will also collect nurse scores for RASS (agitation scores documented as part of usual clinical care), times of scoring and any other delirium or cognitive assessments done as part of usual care (e.g., CAM -ICU, delirium triage screen, mini-cog).

Biosensor data will be coordinated with RASS and presence of delirium using machine learning analysis.

Other data for covariates: medication history/medication administration records, age, gender, length of stay in the ED and in the hospital if applicable. Stage of dementia or most recent cognitive assessment. Baseline skin tone using the expanded Fitzpatrick scale (skin tone scale).

Participant exclusion criteria: patients who are intubated, getting electrical cardioversion or sedation in the ED. Patients who cannot consent due to cognitive impairment and do not have a LAR or caregiver available will also be excluded.

ELIGIBILITY:
Inclusion Criteria:

* adults patients 65+ years old with a known diagnosis of dementia or medical team highly suspects or confirms dementia this visit.
* Emergency Department visit and/or hospitalization anticipated to last >4 more hours from the time of enrollment.

Exclusion Criteria:

* Intubation/mechanical ventilation
* Patients undergoing a procedure requiring sedation
* Patients who cannot consent due to cognitive impairment and do not have a legally authorized representative or caregiver present.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: older adults with dementia in the Emergency Department
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who develop delirium | over the 48 hours of study participation
  The proportion of participants who develop delirium will be determined by one or more positive CAM-ICU 7 (Confusion Assessment Method- Intensive Care Unit 7) assessments during the study participation timeframe. The CAM-ICU 7 is a categorical test with 0 being no delirium and higher numbers signifying different levels of delirium.

SECONDARY OUTCOMES:
Intervention Acceptability | Assessment completed at 48 hours or earlier if discharged prior to 48 hours
  Patient and caregiver acceptability of wearing the biosensor in the hospital will be assessed with a quick 6 question survey based off the Theoretical Framework of Acceptability. Survey questions use likert scales. For example, a score of 1 corresponds to being completely unacceptable and 5 corresponds to being completely acceptable.
Biosensor data usability | 48 hours
  Sometimes wrist biosensors are not able to detect signal well or can be dislodged or removed, which leads to periods of time without usable data. The biosensor data collected from each participant will be assessed for data quality and usability by the statistical analysis team.
Correlation of biosensor array data with clinical delirium | up to 48 hours of biosensor and clinical data per participant
  We will investigate the correlation of the biosensor array data (e.g., heart rate variability, electrodermal activity, and accelerometry) with the development of clinical delirium in the participants. This statistical analysis will be completed asynchronously after all the participants have finished all data collection for the study.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Boyer, MD, Study Director — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No